CLINICAL TRIAL: NCT05474989
Title: LSD Treatment for Persons With Alcohol Use Disorder: A Multicenter, Double-blind, Randomized, Active-placebo Controlled Phase II Study
Brief Title: LSD Treatment for Persons With Alcohol Use Disorder
Acronym: LYSTA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Felix Mueller (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor-Investigator, Felix Mueller, Sponsor-Investigator PD Dr. med. Felix Müller MD, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-00121
Record Dates: First submitted 2022-07-20; First posted 2022-07-26 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Alcohol Use Disorder (AUD)
MeSH Terms: conditions — Alcoholism | interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Subjects in the treatment arm will receive 150 μg LSD (first session) and 150 or 250 μg LSD (second session).
  Interventions: Drug: LSD
- Active placebo (Active Comparator): Subjects in the control arm will receive 10 µg LSD at the first session and 10 µg LSD at the second session.
  Interventions: Drug: Active placebo

INTERVENTIONS:
Drug: LSD — Moderate to high dose LSD
  Arms: Verum
Drug: Active placebo — Low dose LSD
  Arms: Active placebo

SUMMARY:
Alcohol use causes more overall harm than any other drug and is the seventh leading risk factor for both deaths and disability-adjusted life years. Alcohol use disorders (AUD) are among the most common and undertreated mental disorders in developed countries. Pharmacological and psychotherapeutic treatments only show limited efficacy and around 60% of the patients relapse in the short-term after withdrawal.

Lysergic acid diethylamide (LSD) was investigated in numerous clinical trials during the 1950s and 1960s. Specifically, the use of LSD in the treatment of AUD was investigated extensively. A pooled analysis of six historical clinical trials demonstrated, that a single dose of LSD significantly reduced alcohol use at three and six months after LSD administration. However, these trials are limited by several factors, including the use of diagnostic standards that are no longer not up to date, single, high-dose treatment regimes, missing biological assessment for alcohol use, and no consequent assessment of blinding.

Therefore, the present study aims to evaluate the safety and efficacy of LSD for the treatment of AUD and addresses the shortcomings of previous studies. The trial has a double-blind, active placebo-controlled, randomized, parallel design and will be conducted in specialized treatment centers for addictive disorders in Switzerland. The study will include 126 patients after withdrawal treatment and will primarily assess the efficacy of LSD for the treatment of AUD. Patients will be treated using a 1:1 allocation. Each arm will last 20 weeks and will comprise nine study visits without drug administration and two study days involving LSD or active placebo administration. In the first session, patients in the treatment group will receive a dose of 150 µg LSD, followed by another 150 µg or 250 µg LSD in the second session, which will take place approximately 4 weeks after the first session.

The primary outcome is the mean of percent heavy drinking days after administration of two doses of LSD at 3 months follow-up. Additionally, the study will assess neurobiological mechanisms of action and several other measures.

ELIGIBILITY:
Key inclusion criteria:

* age ≥ 25 years
* moderate to severe AUD
* completion of a qualified detoxification for AUD within 30 days prior to screening
* a minimum of 4 heavy drinking days within the last 30 days before detoxification
* intention to stop or decrease drinking

Key exclusion criteria:

* significant alcohol withdrawal symptoms at screening
* participating or starting in any formal treatment for AUD until completion of visit 9
* cognitive impairment
* borderline personality disorder
* current post-traumatic stress disorder
* current suicidality or history of a serious suicide attempt
* significant prodromal symptoms
* history of a diagnosis of a psychotic or bipolar disorder in subjects or first-degree relatives
* pregnancy or breast-feeding
* lack of safe contraception are exclusion criterion for women only

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Percent heavy drinking days | Period of three months after the second intervention
  The primary outcome is the mean of percent heavy drinking days after administration of two doses of LSD assessed with the alcohol timeline follow-back (TLFB) questionnaire compared between treatment groups

SECONDARY OUTCOMES:
Cortical thickness measured with MRI | Two weeks before first administration, two and 12 weeks after second administration
  Changes in the cortical thickness of ACC, PCC, and PFC
The volume of the striatum measured with MRI | Two weeks before first administration, two and 12 weeks after second administration
  Changes in the volume of the striatum
White matter microstructure measured with MRI | Two weeks before first administration, two and 12 weeks after second administration
  Changes in white matter microstructure in the cingulum bundle and the PFC-striatal connection pathway
Days to first heavy drinking day | Three months after the second intervention
  Days to first heavy drinking day after first and second administration assessed with TLFB
Days to first drinking day | Three months after the second intervention
  Days to first drinking day assessed after first and second administration assessed with TLFB
Percent days abstinent | Three months after the second intervention
  Percent days abstinent after first and second administration assessed with TLFB
Drinks per drinking day | Three months after the second intervention
  Drinks per drinking day after first and second administration assessed with TLF
Adverse consequences of alcohol use | Three months after the second intervention
  Adverse consequences of alcohol use assessed with Short Inventory of Problems
Craving | Three months after the second intervention
  Craving assessed with Obsessive Compulsive Drinking Scale
Ethyl glucuronide | Screening and three months after the second intervention
  Ethyl glucuronide (EtG) in hair
Phosphatidylethanol | Screening, day of first intervention, day of second intervention, three months after the second intervention
  Phosphatidylethanol (PEth) in blood
General health | Three months after the second intervention
  General health assessed with General Health Questionnaire
Depression | Three months after the second intervention
  Hamilton Depression Rating Scale
Anxiety | Three months after the second intervention
  Beck Anxiety Inventory
Blinding | In the evening after administration 1 (week 4) and administration 2 (week 8), respectively
  Blinding will be assessed directly after each session by asking patients and therapists to guess the group assignment ("high dose", "low dose", "don't know") and to provide their degree of certainty (using a visual analogue scale) of their guess.
Safety: Adverse events | Week 0 to week 20
  Adverse events will be documented at each visit and each session.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Hospital of Psychiatry, University of Basel, Basel
  - University Hospital of Psychiatry, University of Bern, Bern

IPD SHARING:
Plan to Share IPD: No